CLINICAL TRIAL: NCT02396420
Title: Phase II, Single Center, Single Arm, Open Label Investigation of Prostate Artery Embolization as a Treatment for Benign Prostatic Hyperplasia in Men With Prostates Larger Than 90 Grams
Brief Title: Prostate Artery Embolization as a Treatment for Benign Prostatic Hyperplasia in Men With Prostates Larger Than 90 Grams
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: IP received FDA clearance for use in PAE as treatment for BPH.
Sponsor: South Florida Medical Imaging, PA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAE001
Record Dates: First submitted 2015-03-12; First posted 2015-03-24 (Estimated); Results first posted 2018-11-06 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-10

CONDITIONS: Prostatic Hyperplasia
Keywords: BPH; prostatic hyperplasia; enlarged prostate; benign prostatic hypertrophy
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment arm (Experimental): Patients will receive prostate artery embolization (PAE) with Embosphere Microspheres.
  Interventions: Device: Embosphere Microspheres

INTERVENTIONS:
Device: Embosphere Microspheres

SUMMARY:
The purpose of the study is to evaluate improvement in symptoms related to benign prostatic hyperplasia (BPH) in men treated with prostate artery embolization (PAE) using Embosphere Microspheres.

DETAILED DESCRIPTION:
The study will evaluate improvement in symptoms associated with benign prostatic hyperplasia (BPH) in men with prostates larger than 90 grams treated with prostate artery embolization (PAE). Symptoms will be assessed utilizing the International Prostate Symptom Score (IPSS) to evaluate change from baseline at 12 months post PAE.

ELIGIBILITY:
Inclusion Criteria:

* Patient has provided signed informed consent
* Patient is aged greater than or equal to 40 and less than or equal to 89 years of age
* Patient has a prostate size between 90g and 200g, as determined by MRI
* Patient has experienced lower urinary tract symptoms (LUTS) for at least 6 months prior to study enrollment
* Patient has an IPSS score of at least 13 at baseline
* Patient is either: refractory to medical treatment, contraindicated to medical treatment, OR refuses medical treatment
* Patient either: refuses surgical treatment OR is contraindicated for surgical treatment
* Patient meets ONE of the following criteria: baseline PSA < 4.0ng/mL (no prostate biopsy required) OR baseline PSA >/= 4 ng/mL AND a negative prostate biopsy (minimum 12 core biopsy) within the prior 12 months

Exclusion Criteria:

* History of prostate, bladder, or rectal cancer
* History of transurethral resection of the prostate (TURP), open prostate surgery, or radiofrequency or microwave therapies
* History of open bladder, rectosigmoid colon, or other pelvic surgery
* Patient is unwilling to discontinue alpha blockers 1 month after study treatment
* Patient is unwilling to discontinue 5-alph reductase inhibitors 1 month after study treatment
* Neurogenic bladder or other neurologic disorder impacting bladder function such as Parkinson's disease, multiple sclerosis, cerebral vascular accident or diabetes
* Any other confounding bladder or urethral pathology, including urethral stricture, bladder neck contracture, or bladder atonia
* Active prostatitis or urinary tract infection
* Cystolithiasis within the past 3 months
* Serum creatinine > 1.7mg/dL
* Inability to discontinue oral anticoagulant 2-5 days prior to study treatment
* Coagulation disturbances not normalized by medical treatment
* Iodinated contrast allergy that, in the opinion of the Investigator, cannot be adequately premedicated
* Gelatin allergy
* Known severe peripheral vascular disease or major iliac arterial occlusive disease
* Interest in future fertility
* Clinically significant cardiac arrhythmia or other cardiac disease (including congestive heart failure), uncontrolled diabetes mellitus, clinically significant respiratory disease, or known immunosuppression
* Other condition that the Investigator believes puts the patient at risk for a complication during the procedure

Ages: 40 Years to 89 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-09-24 (Actual); Primary Completion 2016-11-17 (Actual); Study Completion 2016-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rush, MD, Principal Investigator — South Florida Medical Imaging, Holy Cross Hospital
Locations (1):
- Holy Cross Hospital, Fort Lauderdale, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Following FDA and IRB approval for the study, recruitment began and the first subject was enrolled for the study on September 24, 2015. Enrollment was closed on June 29, 2017.
Pre-assignment Details: The study involved a screening period during which patient eligibility was determined. There were no screen failures.
Groups:
- Treatment Arm: Patients will receive prostate artery embolization (PAE) with Embosphere Microspheres.
  Embosphere Microspheres
Period: Overall Study
Arm/Group | Treatment Arm
Started | 2
1 Month Post PAE | 2
3 Months Post PAE | 2
6 Months Post PAE | 2
Completed (12 Months Post PAE) | 1
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment Arm: Prostate artery embolization (PAE) with Embosphere Microspheres.
  Embosphere Microspheres
Arm/Group | Treatment Arm
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 67.5 [66 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2
Use of 5 alpha reductase inhibitors [Count of Participants; unit: Participants] | 1
Use of alpha adrenergic blockers [Count of Participants; unit: Participants] | 2
Use of other medications or supplements [to treat BPH] [Count of Participants; unit: Participants] | 1
Use of other BPH treatments [Count of Participants; unit: Participants] | 0

OUTCOME MEASURES:

1. Primary Outcome: Improvement of Symptoms Associated With Benign Prostatic Hyperplasia (BPH) as Assessed by the International Prostate Symptom Score (IPSS)
Description: The outcome measure was the International Prostate Symptom Score (IPSS). The IPSS is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic). A higher score means a worse outcome.
Time Frame: 12 months
Population: Analysis population includes all subjects in the treatment arm who received unilateral or bilateral prostate artery embolization (PAE) and completed the study thru Visit 5 (12 month follow-up).
Measure: Number; unit: units on a scale
Groups:
- Treatment Arm: This is a single arm study. This arm includes all subjects with study eligibility confirmed during the screening period and Visit 1 (Prostate Artery Embolization) completed within 4 weeks of eligibility confirmation.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 1
units on a scale | 7
Statistical Analysis 1: Comparison: Treatment Arm; Test type: Other; Statistical analysis was not performed as the sample size is insufficient to have confidence that the results would be meaningful for the overall target population

2. Secondary Outcome: Change From Baseline in Prostate Size, as Determined by MRI
Description: Prostate size was determined by measuring the prostate with magnetic resonance imaging (MRI) and calculating length x width x height x pi/6.
Time Frame: Baseline and 12 months
Population: as for outcome 1
Measure: Number; unit: grams
Arm/Group | Treatment Arm
Number analyzed (Participants) | 1
grams | 111
Statistical Analysis 1: Comparison: Treatment Arm; Test type: Other; [other analysis details as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in Peak Urine Flow Rate (Qmax) Determined by Urodynamic Testing
Description: Peak urine flow rate (Qmax) is the greatest volumetric flow rate of urine during urination, measured as the quantity of urine excreted in a specified period of time (per second or per minute). Qmax has become a primary objective parameter of treatment outcomes for various surgical and medical therapies for BPH. Unlike other prominent parameters of treatment outcome, Qmax responds minimally to placebo, making it an objective tool when evaluating a patient's response to therapy.
Time Frame: 12 Months
Population: The one subject who completed the study thru Visit 5 refused to undergo urodynamic testing at Visit 5. As a result the Qmax was not obtained. This was reported as a protocol deviation in the study.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 0
Statistical Analysis 1: Comparison: Treatment Arm; Test type: Other; [other analysis details as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline in Post Void Residual Volume (PVR) as Determined by Urodynamic Testing
Description: Post void residual is a measurement of the amount of urine left in the bladder after voiding. It has traditionally been used to evaluate efficacy of treatment efforts. A positive response to treatment is associated with decreased PVR volumes.
Time Frame: 12 Months
Population: The one subject who completed the study thru Visit 5 refused to undergo urodynamic testing at Visit 5. As a result the PVR was not obtained. This was reported as a protocol deviation in the study.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 0
Statistical Analysis 1: Comparison: Treatment Arm; Statistical analysis was not performed as this data was not available for any subjects in the analysis population; Test type: Other — Statistical analysis was not performed as this data was not available for any subjects in the analysis population; Statistical analysis was not performed as this data was not available for any subjects in the analysis population

5. Secondary Outcome: Change From Baseline in Detrusor Muscle Pressure (Pdet) as Determined by Urodynamic Testing
Description: Detrusor muscle pressure (Pdet) is important when evaluating how strong the detrusor force must be to initiate urine flow in bladder outlet obstruction. Lower Pdet values are associated with a positive response to treatment.
Time Frame: 12 Months
Population: The one subject who completed the study thru Visit 5 refused to undergo urodynamic testing at Visit 5. As a result the Pdet was not obtained. This was reported as a protocol deviation in the study.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 0
Statistical Analysis 1: Comparison: Treatment Arm; Statistical analysis was not performed as this data was not available for any subjects in the analysis population; Test type: Other — Statistical analysis was not performed as this data was not available for any subjects in the analysis population; Statistical analysis was not performed as this data was not available for any subjects in the analysis population

6. Secondary Outcome: Change From Baseline in Erectile Function as Determined by the International Index of Erectile Function (IIEF)
Description: The outcome measure was the International Index of Erectile Function (IIEF). The 15 question IIEF Questionnaire is a validated, multi-dimensional, self-administered investigation found to be useful in the clinical assessment of erectile dysfunction and treatment. It is examines the four main domains of male sexual function: erectile function, orgasmic function, sexual desire, and intercourse satisfaction. The answer to each question is given a score between 0 and 5 for a total score of 0-75 (higher score = less dysfunction). Higher scores mean better outcome.
Time Frame: 12 Months
Population: as for outcome 1
Measure: Number; unit: units on scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 1
units on scale | 69
Statistical Analysis 1: Comparison: Treatment Arm; Test type: Other; [other analysis details as in outcome 1, analysis 1]

7. Secondary Outcome: Change From Baseline in Serum Prostate Specific Antigen (PSA)
Description: Serum prostate specific antigen (PSA) trends over time, may help to improve the specificity of PSA testing in men with BPH. A strong correlation has been demonstrated between prostate volume and serum PSA levels.
Time Frame: Baseline and12 Months
Population: as for outcome 1
Measure: Number; unit: ng/mL
Arm/Group | Treatment Arm
Number analyzed (Participants) | 1
ng/mL | 2.26
Statistical Analysis 1: Comparison: Treatment Arm; Test type: Other; [other analysis details as in outcome 1, analysis 1]

8. Secondary Outcome: Prostate Artery Embolization (PSA) Related Adverse Events
Description: Number of occurrences of adverse events with some relationship to the study procedure or study device. An adverse event (AE) is any untoward medical occurrence in a clinical investigation subject and does not necessarily have to have a causal relationship with the treatment. In order to capture the most potentially relevant safety information during the study, AEs were assessed at each visit. AEs occurring during the clinical trial and the protocol-defined 12-month follow-up period were reported.
Time Frame: 12 Months
Population: Analysis population includes all subjects, in the treatment arm, for whom prostate artery embolization (PAE) was attempted regardless of whether the subject received a unilateral PAE, bilateral PAE, or the attempted PAE was aborted.
Measure: Count of Units; unit: occurrence
Units Other Than Participants: occurrence
Groups:
- Treatment: This is a single arm study. This arm includes all subjects with study eligibility confirmed during the screening period and Visit 1 (Prostate Artery Embolization) completed within 4 weeks of eligibility confirmation.
Arm/Group | Treatment
Number analyzed (Participants) | 2
Number analyzed (occurrence) | 5
occurrence
  Catheter site burning | 1
  Pelvic pain | 1
  Dysuria | 1
  Pollakiuria | 1
  Bladder irritation | 1
Statistical Analysis 1: Comparison: Treatment; Test type: Other; [other analysis details as in outcome 1, analysis 1]

9. Secondary Outcome: Overall Adverse Events
Description: All adverse events will be assessed for severity, relationship to study treatment, subsequent treatment required, and outcome
Time Frame: 12 Months
Population: as for outcome 8
Measure: Number; unit: occurrence
Arm/Group | Treatment
Number analyzed (Participants) | 2
occurrence
  Catheter site burning | 1
  Pelvic pain | 1
  Dysuria | 1
  Pollakiuria | 1
  Bladder irritation | 1
  Nasopharyngitis | 1
  Urinary tract infection | 2
  Acute myocardial infarction | 1
  Acute sinusitis | 1
  Allergic rhinitis | 1
Statistical Analysis 1: Comparison: Treatment; Test type: Other; [other analysis details as in outcome 1, analysis 1]

10. Other Pre Specified Outcome: Total PAE Procedure Time
Description: Parameter measured during the PAE (index procedure) for informational purposes. Total PAE procedure time was defined as time of femoral artery puncture to the time of time sheath removed from femoral artery.
Time Frame: Study treatment hospitalization (expected to be less than 1 day)
Population: as for outcome 8
Measure: Mean (Full Range); unit: minutes
Arm/Group | Treatment Arm
Number analyzed (Participants) | 2
minutes | 179 [130 to 228]
Statistical Analysis 1: Comparison: Treatment Arm; Test type: Other; [other analysis details as in outcome 1, analysis 1]

11. Other Pre Specified Outcome: Total Fluoroscopy Time for PAE
Description: Parameter to be measured during PAE procedure, for informational purposes.
Time Frame: Study treatment hospitalization (expected to be less than 1 day)
Population: as for outcome 8
Measure: Mean (Full Range); unit: minutes
Arm/Group | Treatment
Number analyzed (Participants) | 2
minutes | 60.5 [44 to 77]
Statistical Analysis 1: Comparison: Treatment; Test type: Other; [other analysis details as in outcome 1, analysis 1]

12. Other Pre Specified Outcome: Type of Contrast Media Delivered for PAE
Description: Parameter to be measured during PAE procedure, for informational purposes
Time Frame: Study treatment hospitalization (expected to be less than 1 day)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 2
Participants
  Isovue 370 | 2
  Isovue 300 | 0
Statistical Analysis 1: Comparison: Treatment; Test type: Other; [other analysis details as in outcome 1, analysis 1]

13. Other Pre Specified Outcome: Volume of Contrast Delivered for PAE
Description: Parameter to be measured during PAE procedure, for informational purposes
Time Frame: Study treatment hospitalization (expected to be less than 1 day)
Population: as for outcome 8
Measure: Mean (Full Range); unit: milliliter
Arm/Group | Treatment
Number analyzed (Participants) | 2
milliliter | 160 [60 to 260]
Statistical Analysis 1: Comparison: Treatment; Test type: Other; [other analysis details as in outcome 1, analysis 1]

14. Other Pre Specified Outcome: Volume of Embolic Delivered for PAE
Description: Parameter to be measured during PAE procedure, for informational purposes
Time Frame: Study treatment hospitalization (expected to be less than 1 day)
Population: Analysis population includes all subjects in the treatment arm who received unilateral or bilateral prostate artery embolization (PAE).
Measure: Mean (Full Range); unit: milliliter
Arm/Group | Treatment
Number analyzed (Participants) | 2
milliliter | 8.3 [5.1 to 11.2]
Statistical Analysis 1: Comparison: Treatment; Test type: Other; [other analysis details as in outcome 1, analysis 1]

15. Other Pre Specified Outcome: Number of Origins of Prostatic Blood Supply
Description: Parameter to be measured during PAE procedure, for informational purposes
Time Frame: Study treatment hospitalization (expected to be less than 1 day)
Population: as for outcome 14
Measure: Mean (Full Range); unit: number of vessels
Arm/Group | Treatment
Number analyzed (Participants) | 2
number of vessels
  Origins of blood supply right side: number analyzed (Participants) | 1
  Origins of blood supply right side | 1 [1 to 1]
  Origins of blood supply left side | 1 [1 to 1]
Statistical Analysis 1: Comparison: Treatment; Test type: Other; [other analysis details as in outcome 1, analysis 1]

16. Other Pre Specified Outcome: Duration of Hospitalization Post PAE
Description: Parameter to be measured during PAE procedure, for informational purposes
Time Frame: Study treatment hospitalization (expected to be less than 1 day)
Population: as for outcome 8
Measure: Mean (Full Range); unit: minutes
Arm/Group | Treatment
Number analyzed (Participants) | 2
minutes | 1872 [1869 to 1875]
Statistical Analysis 1: Comparison: Treatment; Test type: Other; [other analysis details as in outcome 1, analysis 1]

17. Other Pre Specified Outcome: Duration of [Urinary] Catheterization Post PAE
Description: Parameter to be measured during PAE procedure, for informational purposes
Time Frame: Study treatment hospitalization (expected to be less than 1 day)
Population: as for outcome 8
Measure: Mean (Full Range); unit: minutes
Arm/Group | Treatment
Number analyzed (Participants) | 2
minutes | 1406 [1390 to 1422]
Statistical Analysis 1: Comparison: Treatment; Test type: Other; [other analysis details as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) occurring during the clinical trial and the protocol-defined 12-month follow-up period were recorded.
Groups:
- Treatment: This is a single arm study. All subjects with eligibility confirmed during the screening period and completing Visit 1 (Prostate Artery Embolization) within 4 weeks of screening are included in the arm.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 1/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=2)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=2)
Catheter site burning (General disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Bladder irritation (Renal and urinary disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2)
Acute sinusitis (Infections and infestations) | 1 (1)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Enrollment was limited due to early study termination. This was a result of Embosphere Microspheres (investigational product for this IDE) receiving FDA clearance for embolization of prostatic arteries for symptomatic benign prostatic hyperplasia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes